CLINICAL TRIAL: NCT04303702
Title: Role of Oxytocin in the Second Stage of Labor: a Randomized Controlled Trial (The ROSSoL Trial)
Brief Title: The Role of Oxytocin in the Second Stage of Labor
Acronym: ROSSoL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: University of Michigan (Other)
Responsible Party: Principal Investigator, Nandini Raghuraman, Assistant Professor, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 201909112
Record Dates: First submitted 2020-03-06; First posted 2020-03-11 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Labor Complication
MeSH Terms: conditions — Obstetric Labor Complications

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Discontinue Oxytocin (Other)
  Interventions: Other: Discontinue Oxytocin
- Continue Oxytocin (Active Comparator)
  Interventions: Drug: Continue Oxytocin

INTERVENTIONS:
Drug: Continue Oxytocin — The administration and titration of oxytocin for labor augmentation is per a hospital based protocol. To summarize, oxytocin is initiated intravenously at 2 milliunits/minute and increased by 2 milliunits/minute every 20 minutes until an adequate contraction pattern is attained or a maximum of 40 millunits/minute has been achieved. This protocol for titration and administration will be applied in this study to the oxytocin group. The intravenous pumps on Labor and Delivery have automated functions for intravenous administration of oxytocin that is milliunit-based and the same routine pumps will be used in this study. The study bag will be administered per current oxytocin protocol. Since patients will already be on oxytocin at time of randomization, their current bag of oxytocin will be continued by the primary provider at a rate of their discretion.
  Arms: Continue Oxytocin
Other: Discontinue Oxytocin — Patients will have their oxytocin discontinued in the second stage of labor. The patient will receive routine maintenance IV fluids per the discretion of the provider.
  Arms: Discontinue Oxytocin

SUMMARY:
This is a randomized controlled trial investigating the utility of oxytocin administration in the second stage of labor.

DETAILED DESCRIPTION:
Oxytocin is widely used on Labor and Delivery units throughout the world.Laboring patients are most likely to initiate oxytocin in the first stage of labor. Among those who receive oxytocin, first stage initiation is far more common than second stage initiation. The goal of first stage administration is to increase uterine contractility and cause cervical dilation, particularly in patients who have epidural analgesia. Once complete cervical dilation has been achieved, most providers choose to continue oxytocin in the second stage of labor for the theoretic benefit of increased expulsion "power" while pushing. This practice is currently not evidence-based as the limited data thus far suggests no difference in operative deliveries with the use of oxytocin augmentation in general. The benefits and risk of oxytocin continuation in the second stage of labor is unknown. Oxytocin administration is associated with the risk of uterine tachysystole, postpartum hemorrhage,and maternal hyponatremia. These risks call for a closer look at prolonged oxytocin use past the first stage of labor. This is a randomized controlled trial investigating the utility of oxytocin administration in the second stage of labor.

ELIGIBILITY:
Inclusion Criteria:

* Nulliparous pregnant women >/= 37 weeks gestation
* Singleton pregnancies
* Admission for induction of labor or spontaneous labor

Exclusion Criteria:

* Multiple gestations
* Multiparous patients
* Patients with major fetal anomalies
* Not on oxytocin at the time of complete cervical dilation
* Patients with fetal head visible at the perineum on diagnosis of complete cervical dilation
* Maternal medical condition that prohibits prolonged second stage

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Second stage duration | During admission for delivery
  Time interval from complete cervical dilation to delivery of fetus

SECONDARY OUTCOMES:
Rate of operative delivery | During admision for delivery
  Rate of cesarean section and operative vaginal delivery including forcep or vacuum
Rate of Postpartum hemorrhage | During admission for delivery
  Estimated blood loss >500 mL for vaginal delivery and >1000 mL for cesarean delivery
Estimated blood loss | During admission for delivery
  Estimated blood loss at time of delivery (mL)
Rate of chorioamnionitis during the second stage of labor | During admission for delivery
  Chorioamnionitis diagnosed at discretion of primary provider during the second stage of labor
Rate of endometritis | During admission for delivery
  Postpartum endometritis as diagnosed by primary provider
Rate of severe perineal laceration | During admission for delivery
  3rd or 4th degree perineal laceration
Rate of composite neonatal morbidity | During admission for delivery
  1 or more of the following: death, birth injury, umbilical artery acidosis, respiratory distress, transient tachypnea, meconium aspiration with pulmonary hypertension, hypoxic-ischemic encephalopathy, hypoglycemia, hypothermia treatment, or suspected neonatal sepsis.

CONTACTS AND LOCATIONS:
Locations (1):
- Barnes Jewish Hospital, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Undecided